CLINICAL TRIAL: NCT05528705
Title: A Randomized, Parallel-group, Placebo-controlled, Single-blind, Investigator Initiated Trial to Evaluate Efficacy and Safety of LAENNEC (Human Placenta Hydrolysate) Administered by Ultrasonography Guided Subacromial Bursa Injection in Patients With Shoulder Impingement Syndrome
Brief Title: Investigator Initiated Trial to Evaluate Efficacy and Safety of LAENNEC (Human Placenta Hydrolysate) Administered by Ultrasonography Guided Subacromial Bursa Injection in Patients With Shoulder Impingement Syndrome
Acronym: PAIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Green Cross Wellbeing (Industry)
Collaborators: Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: LAEN-PAIN
Record Dates: First submitted 2022-09-01; First posted 2022-09-06 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Shoulder Impingement Syndrome
MeSH Terms: conditions — Shoulder Impingement Syndrome | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LAENNEC (Experimental): 4ml once a week for 3 weeks of Subacromial spatial administration + conservative treatment
  Interventions: Biological: LAENNEC
- 0.9% Normal saline (Active Comparator): 4ml once a week for 3 weeks of Subacromial spatial administration + conservative treatment
  Interventions: Other: 0.9% normal saline

INTERVENTIONS:
Biological: LAENNEC — Subacromial spatial administration
  Other Names: Human Placenta Hydrolysate
  Arms: LAENNEC
Other: 0.9% normal saline — Subacromial spatial administration
  Arms: 0.9% Normal saline

SUMMARY:
To patients with shoulder collision syndrome, LAENNEC (Human Placenta Hydrolysate) is administered as an injection in the ultrasonic induction underglone, to evaluate the effectiveness and safety.

ELIGIBILITY:
Inclusion Criteria:

1. At the time of screening, 19 or 70 years
2. Those who are suspected of rotator cuff lesions or damage due to shoulder pain
3. Those who are judged to have a shoulder joint disease during screening
4. Neer test, Hawkins-Kennedy inspection, job test, Painful Arc inspection or resisted showder external rotation test
5. Those with a significant pain of 30 mm of Visual Analogue Scale (VAS)
6. Those who can sign a test subject or to comply with the matters required for clinical trials.

Exclusion Criteria:

1. A person who appears in the movement of two or more shoulder joints with more than 50% of the joint movement limit on the passive shoulder joint operation scope test.
2. Those who have confirmed the rupture of the entire layer by ultrasound
3. Those with serious damage to the shoulders and the past power
4. Those who have suspected fractures, dislocations, degenerative arthritis, and calcification in the shoulder radiation test in the shoulder radiation test.
5. Those who complain of shoulder pain due to stroke, spinal cord injury, and other surgery
6. Those with other shoulder diseases other than fifty dogs (rheumatoid arthritis, osteoarthritis, bone defect injuries, malignant tumors, etc.)
7. Those who are accompanied by diseases of cervical spine or other upper limbs that have a significant effect on the shoulder
8. Those who have performed steroid injections in the joint steel within 3 months of participation in clinical trials
9. Those who have administered anti -inflammatory drugs within two weeks of participation in clinical trials
10. Those with all other joint diseases that have musculoskeletal diseases that may affect effective evaluation, or that it is impossible to participate in this clinical trial.
11. Those who are diagnosed with mental illness and taking drugs
12. Pregnant women and lactation departments, fertility women who are not willing to contraceptive during the clinical trial period
13. Those who have received medication, oriental medicine, physical therapy, and injection treatment in relation to shoulder pain within the last two weeks 14 Those who are participating in other clinical trials during screening

15. Those who determine that other testors are inadequate

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2022-09-13 (Actual); Primary Completion 2023-10-23 (Actual); Study Completion 2024-01-31 (Actual)

PRIMARY OUTCOMES:
Change amoust of VAS (visual analogue scale) | week 0 and 12

SECONDARY OUTCOMES:
Change amoust of VAS (visual analogue scale) | week 1, 2, 3 and 6
Change amoust of SPADI | week 1, 2, 3, 6 and 12
Change amoust of EQ-5D-5L | week 1, 2, 3, 6 and 12

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Keimyung University Dongsan Hospital, Daegu
  - Chung-Ang University Gwangmyeong Hospital, Gwangmyeong
  - Chung-Ang University Hospital, Seoul

REFERENCES:
- [Derived] Kim DH, Park MW, Shin HI, Lee BC, Kim DK, Cho CH, Kim YJ. Effectiveness and safety of human placenta hydrolysate injection into subacromial space in patients with shoulder impingement syndrome: a single-blind, randomized trial. BMC Musculoskelet Disord. 2025 Jan 3;26(1):11. doi: 10.1186/s12891-024-08266-4. PMID 39754114